CLINICAL TRIAL: NCT01536782
Title: The Optimal Tube Feeding Method in Head and Neck Cancer Patients: A Comparison Between Bolus, Gravity, and Tube Feeding Pump.
Brief Title: Optimal Tube Feeding Method in Head and Neck Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the company
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012-026
Record Dates: First submitted 2012-01-23; First posted 2012-02-22 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; chemoradiation therapy; bolus feeding; gravity feeding; pump feeding; optimal enteral feeding method; To determine the optimal tube feeding method by analyzing percent weigtht loss.; To determine the optimal tube feeding method by analyzing tolerance of enteral feeds.; To determine the optimal tube feeding method by analyzing percent met of estimated calories and protein.
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — NOP-bolus regimen; Gravitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bolus (Active Comparator): Upon tube feeding initiation determined by the HNC multidisciplinary team, the patients will be randomized into three different groups, each consisting of 20 patients each: Bolus (Group 1), Gravity (Group 2), and Pump (Group 3). The randomization process within these three groups will based on 1) age and 2) estimated caloric need. For example, if we have three 60-year-old patients whose estimated kcals needs are ≤ 1900kcals/day, then each patient will be randomized to either Bolus, Gravity or Pump group. Another example is that if we have two 45-year-old patients whose estimated needs are 2400kcals/day, then one patient will randomly be assigned to the Bolus group, and the other one will be randomly assigned to the Gravity group. The third patient that will fit that category will be assigned to the Pump group.
  Interventions: Procedure: Bolus
- Gravity (Active Comparator): Upon tube feeding initiation determined by the HNC multidisciplinary team, the patients will be randomized into three different groups, each consisting of 20 patients each: Bolus (Group 1), Gravity (Group 2), and Pump (Group 3). The randomization process within these three groups will based on 1) age and 2) estimated caloric need. For example, if we have three 60-year-old patients whose estimated kcals needs are ≤ 1900kcals/day, then each patient will be randomized to either Bolus, Gravity or Pump group. Another example is that if we have two 45-year-old patients whose estimated needs are 2400kcals/day, then one patient will randomly be assigned to the Bolus group, and the other one will be randomly assigned to the Gravity group. The third patient that will fit that category will be assigned to the Pump group.
  Interventions: Procedure: Gravity
- Pump (Active Comparator): Upon tube feeding initiation determined by the HNC multidisciplinary team, the patients will be randomized into three different groups, each consisting of 20 patients each: Bolus (Group 1), Gravity (Group 2), and Pump (Group 3). The randomization process within these three groups will based on 1) age and 2) estimated caloric need. For example, if we have three 60-year-old patients whose estimated kcals needs are ≤ 1900kcals/day, then each patient will be randomized to either Bolus, Gravity or Pump group. Another example is that if we have two 45-year-old patients whose estimated needs are 2400kcals/day, then one patient will randomly be assigned to the Bolus group, and the other one will be randomly assigned to the Gravity group. The third patient that will fit that category will be assigned to the Pump group.
  Interventions: Device: Pump

INTERVENTIONS:
Procedure: Bolus — The patients will be randomized into 3 different groups: Bolus, Gravity, and Pump. The randomization process will be based on age and estimated caloric needs (i.e if we have three 60-year-old patients whose estimated kcals needs are ≤ 1900kcals/day, then each patient will be randomized to either of the groups).
  Each patient from each group will be receiving tube feeding education to their by RD. For consistency reasons, the same type of tube feeding formula (1.5 kcal/ml, no fiber) will be used. Patients' weight, tube feeding tolerance, and amount of estimated calories and protein met will be monitored weekly.
  Arms: Bolus
Procedure: Gravity — The patients will be randomized into 3 different groups: Bolus, Gravity, and Pump. The randomization process will be based on age and estimated caloric needs (i.e if we have three 60-year-old patients whose estimated kcals needs are ≤ 1900kcals/day, then each patient will be randomized to either of the groups).
  Each patient from each group will be receiving tube feeding education to their by RD. For consistency reasons, the same type of tube feeding formula (1.5 kcal/ml, no fiber) will be used. Patients' weight, tube feeding tolerance, and amount of estimated calories and protein met will be monitored weekly.
  Arms: Gravity
Device: Pump — The patients will be randomized into 3 different groups: Bolus, Gravity, and Pump. The randomization process will be based on age and estimated caloric needs (i.e if we have three 60-year-old patients whose estimated kcals needs are ≤ 1900kcals/day, then each patient will be randomized to either of the groups).
  Each patient from each group will be receiving tube feeding education to their by RD. For consistency reasons, the same type of tube feeding formula (1.5 kcal/ml, no fiber) will be used. Patients' weight, tube feeding tolerance, and amount of estimated calories and protein met will be monitored weekly.
  Arms: Pump

SUMMARY:
The purpose of this study is to assess the optimal tube feeding method (bolus, gravity or pump) by analyzing percent weight loss, tolerance of enteral feeds, and percent of estimated calorie and protein needs in 60 patients with squamous cell carcinoma of the head and neck undergoing chemoradiation therapy.

DETAILED DESCRIPTION:
It is a great challenge to maintain the nutritional status of the head and neck cancer (HNC) patients through treatment advances such as combined chemoradiation therapy or CRT. For all these reasons, HNC patients undergoing treatment, frequently require alternate methods of nutrition support such as as enteral tube feeding via a gastrostomy tube.Upon gastric tube feeding initiation, the registered dietitian (RD) must consider the three different methods: bolus (using a syringe), gravity (using gravity feeding bags), and pump (using a tube feeding pump).

Typically, patients are started on bolus (OPTION A), changed to gravity (OPTION B) if bolus feeds are not tolerated, and ultimately changed to pump (OPTION C) if gravity feeds are not tolerated. The concern is that in this process of starting with OPTION A, and moving to OPTION B or further to OPTION C, the patient may experience unintentional weight loss and dehydration related to tube feeding intolerance and/or tube feeding inadequacy. Consequently, this places the patient at risk of, but not limited to, hospital admission for dehydration and/or malnutrition, and treatment interruption. Therefore, exploring the idea of an optimal feeding method and starting patients on it from the beginning, may improve patient outcomes in terms of nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 18 years or older
* Diagnosis of SCCHN undergoing concurrent chemoradiation therapy (including patients who received induction therapy upfront

Exclusion Criteria:

* Patients who have a small bowel feeding tube (only tube feeding via pump is allowed in this case)
* Patients with history of gastric surgery which may have resulted in altered gastrointestinal function
* Patients with history of uncontrolled diabetes and/or gastroparesis which may interfere with gastric emptying and inability to tolerate bolus feeds
* Patients at high risk of aspiration in which case slower feeds by using gravity or pump are indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
percent weight loss | 2 years
tolerance of enteral feedings | 2 Years

SECONDARY OUTCOMES:
Percent met of estimated calories and proteins | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andreea Nguyen, MS in Nutrition, Principal Investigator — Baylor Health Care System
Locations (1):
- Charles A. Sammons Cancer Center at Baylor University Medical Center, Dallas, Texas, United States